CLINICAL TRIAL: NCT02256280
Title: Decurarization After Thoracic Anesthesia - A Prospective Multicenter Double-blind Randomized Trial Comparing Sugammadex vs Neostigmine Reversal After Thoracic Anesthesia
Brief Title: A Randomized Double Blind Controlled Trial Comparing Sugammadex and Neostigmine After Thoracic Anesthesia
Acronym: DATA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low recruiting rate due to not activation of some collaborator centers
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Principal Investigator, Federico Piccioni, MD, Principal Investigator, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: INT-91/14; 2014-002021-35 (EudraCT Number)
Record Dates: First submitted 2014-09-24; First posted 2014-10-03 (Estimated); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Neuromuscular Blockade
Keywords: Neuromuscular blockade; Thoracic surgery
MeSH Terms: interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- S Group (Experimental): Sugammadex 2 or 4 mg/kg iv once at the end of surgery
  Interventions: Drug: Sugammadex
- N Group (Active Comparator): Neostigmine 0.05 or 0.07 mg/kg (+ atropine 0.02 mg/kg) iv once at the end of surgery
  Interventions: Drug: Neostigmine

INTERVENTIONS:
Drug: Sugammadex — Sugammadex will be diluted in a saline water solution in a 10 mL syringe.
  Administration will be according to the neuromuscular blockade:
  * If Post tetanic count = 1-15: 4 mg/kg
  * If at least 1 twitch at the Train-of-four stimulation: 2 mg/kg
  Other Names: Bridion
  Arms: S Group
Drug: Neostigmine — Neostigmine will be diluted with atropine in a saline water solution in a 10 mL syringe.
  Administration will be according to the neuromuscular blockade:
  * If Post tetanic count = 1-15: 0.07 mg/kg
  * If at least 1 twitch at the Train-of-four stimulation: 0.05 mg/kg Atropine will be administered at a 0.02 mg/kg dosage.
  Other Names: Intrastigmina
  Arms: N Group

SUMMARY:
At the end of anesthesia it's important to avoid residual neuromuscular block to ensure adequate respiratory function preventing postoperative pulmonary complications. This trial compares the neuromuscular block reversal with different drugs (sugammadex vs neostigmine) after thoracic anesthesia. The trial main objective is to demonstrate that sugammadex is faster than neostigmine to reach a Train-of-four-Ratio (TOF-ratio) of 0.9 after thoracic anesthesia, demonstrating that sugammadex allows a faster extubation. Other main purpose is to verify if there is a difference between sugammadex and neostigmine as regards adverse events after extubation and in the postoperative period (until the 30th day after surgery).

Note: TOF-ratio is defined as the ratio of the fourth muscular twitch/first twitch value during an accelerometric train-of-four stimulation.

DETAILED DESCRIPTION:
Patients undergoing thoracic surgery will receive rocuronium as neuromuscular blocking agent. Anesthesia and neuromuscular blockade will be managed freely until the end of surgery. Then patients will be randomized to receive intravenous sugammadex or neostigmine/atropine as follows:

Sugammadex group:

* If Post tetanic count (PTC)=1-15: sugammadex 4 mg/kg
* If at least 1 twitch at the Train-of-four stimulation: sugammadex 2 mg/kg

Neostigmine group:

* If PTC=1-15: neostigmine 0.07 mg/kg + atropine 0.02 mg/kg
* If at least 1 twitch at the Train-of-four (TOF) stimulation: neostigmine 0.07 mg/kg + atropine 0.02 mg/kg

ELIGIBILITY:
Inclusion Criteria:

* Subjects scheduled for pulmonary resection, lobectomy, pneumonectomy, bullectomy, pleurodesis
* Age 18-70 years
* American Society of Anesthesiologists (ASA) class 1, 2, 3
* Body mass Index (BMI) = 18-30 kg/m2

Exclusion Criteria:

* Subjects scheduled for esophagectomy, thoracectomy, vascular resection
* Chronic Obstructive Pulmonary Disease (COPD) Gold class III e IV, respiratory infection, asthma
* Preoperative Forced Expiratory Volume in 1 second (FEV1) < 60% of predicted, Forced Expiratory Volume in 1 second/Forced Vital Capacity ratio (FEV1/FVC) <70%
* Preoperative Diffusion Lung capacity for carbon monoxide/Alveolar Volume ratio (DLCO/VA) < 60% of predicted
* Preoperative oxygen saturation (SpO2) <92% or Partial pressure of oxygen in arterial blood/Fraction of inspired oxygen (PaO2/FiO2) ratio <300
* Cardiovascular disease with Metabolic Equivalent of Tasks (METS) score less than 4
* Neuromuscular disorder
* Kidney failure defined as Estimated Glomerular Filtration Rate (eGFR) < 30 ml/min/1,73 m2
* Pregnant women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Mean time from reversal administration to Train-of-four-ratio (TOF-ratio) = 0.9 | At the end of general anesthesia
  Time from reversal administration to at least 3 TOF-ratio value = or > 0.9

SECONDARY OUTCOMES:
Mean time from reversal administration to TOF-ratio = 1.0 | At the end of general anesthesia
  Time from reversal administration to at least 3 TOF-ratio value = or > 1.0
Mean time from reversal administration to extubation | At the end of anesthesia
  Time from reversal administration to tracheal extubation
Muscular weakness incidence | In the first 60 minutes after extubation
  Measured by the tongue depressor test
Hypoxemia or hypercapnia incidence | In the first 60 minutes after extubation
  Hypoxemia defined as Partial pressure of oxygen in arterial blood/Fraction of inspired oxygen ratio (PaO2/FiO2) < 300. Hypercapnia defined as Partial pressure of carbon dioxide in arterial blood (PaCO2) > 45 mmHg.
Adverse events incidence | In the first 60 minutes after extubation
  Incidence of nausea or vomit, abdominal pain, cardiac arrhythmias, hypotension coded according to the Medical Dictionary for Regulatory Activities (MedDRA) terminology
Postoperative complications incidence | Participants will be followed for the duration of hospital stay, an expected average of 7 days
  Incidence of medical and surgical complications coded according to the MedDRA terminology

OTHER OUTCOMES:
Mean time of hospital discharge | Participants will be followed for the duration of hospital stay, an expected average of 7 days
  Time from intervention date to the hospital discharge
Postoperative complications incidence | At 30 days after surgery
  Incidence of medical and surgical complications coded according to the MedDRA terminology

CONTACTS AND LOCATIONS:
Overall Officials: Federico Piccioni, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Mi, Italy